CLINICAL TRIAL: NCT05891431
Title: Acceptability and Preliminary Effectiveness of a Mobile Health Intervention (Untire App) for Adult Cancer Patients and Survivors With Cancer Related Fatigue: A Pilot Clinical Study
Brief Title: Engagement and Acceptability of the Untire mHealth App
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Tired of Cancer B.V. (Industry)
Responsible Party: Principal Investigator, Emil Vuillermoz, Principle Investigator, University of Bath
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 318755
Record Dates: First submitted 2023-05-06; First posted 2023-06-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer-related Problem/Condition; Cancer-related Fatigue
Keywords: Cancer; mHealth; Fatigue; app; self-management; engagement; Acceptability; Quality of life
MeSH Terms: conditions — Neoplasms; Fatigue; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A within groups study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Untire app (Experimental): Participants will be given access to the Untire app.
  Untire is a mHealth app and a registered medical device (ICD10 code R53.83 Fatigue) introduced in 2018 to treat Cancer Related Fatigue in adults.
  Interventions: Device: Untire mobile app

INTERVENTIONS:
Device: Untire mobile app — The Untire app is an mHealth intervention (digitally delivered using a smartphone app).
  Untire offers a comprehensive program to help you understand cancer fatigue and gives a physical activity program, stress reduction exercises and tips to manage your energy level.

SUMMARY:
The aim of this study will be to assess the engagement and acceptability of the Untire mHealth intervention for adults with cancer related fatigue. Acceptability will be assessed after 2, 4, 6 and 12 weeks of app use. Participants (both those competed the study and those who stopped using the app) will be asked about their engagement with the app.

A secondary aim of this study will be to provide preliminary efficacy outcomes of the Untire intervention in reducing fatigue and QoL in adults experiencing cancer related fatigue.

DETAILED DESCRIPTION:
Cancer-related fatigue (CRF) is one of the most severe and commonly reported side effects of cancer treatment. There is a growing body of evidence that mHealth interventions (digitally delivered using a smart phone app) are effective at reducing CRF. The Untire app is a mHealth app is a registered medical device (ICD10 code R53.83 Fatigue) introduced in 2018 to treat CRF. One limitation common to most digitally delivered interventions is high levels of study drop out and decreased app use over time.

The aim of this study will be to assess the engagement and acceptability of the Untire mHealth intervention for adults with cancer related fatigue.A secondary aim of this study will be to provide preliminary efficacy outcomes of the Untire intervention in reducing fatigue and QoL in adults experiencing cancer related fatigue. The hypotheses for these efficacy outcomes are:

Hypothesis 1: Participants using the Untire app intervention will show reduced levels fatigue (as measured by scores on the fatigue subscale of the FACT-F) after 12 weeks compared to baseline.

Hypothesis 2: Participants using the Untire app intervention will show improved QoL (as measured by scores on the FACT-F) after 12 weeks compared to baseline.

Design:

A within groups study design will be used to evaluate the acceptability, engagement, and preliminary efficacy of the Untire mHealth intervention in adults with cancer related fatigue.

Participants:

Participants will be recruited through the following channels:

* NHS Cancer Treatment centres within the South West of England.
* Charities and third sector organisations: Youth Cancer Trust, Cancer Support UK, Macmillan, Shine.
* Social media: support groups/ networks on Facebook and Instagram: Cancer Awareness for Teens and Twenties (CATTs).

Engagement will be measured through retention and adherence rates over 12-week and in app use data; duration of app use and time spent on each activity within the app. Acceptability will be measured using the Acceptability E-scale and Digital Working Alliance Inventory collected at each time point. Other measures will include The Functional Assessment of Chronic Illness Therapy - Fatigue (FACT-F) to provide preliminary data on effectiveness. The investigators also aim to contact participants who stop using the app or drop out of the study. This will be via email or telephone so they can provide qualitative feedback on the app.

Rationale:

The aim of looking at user engagement and acceptability was chosen as this is an area that is less well studied in mHealth interventions. Improving user engagement can be clinically significant as it can increase the amount of time patients spend using the intervention leading to better health outcomes. Looking at levels of acceptability and engagement across our sample will help us identify whether sample characteristics (such as age of user, cancer type) impact acceptability or engagement. This along with user feedback will help us to develop and tailor the Untire intervention to better fit with specific patient groups. Following up participants who have stopped using the app is something that is not normally possible in larger randomised control trials and will hopefully provide useful data on acceptability which can be used to develop the intervention in the future.

The study protocol has been developed with the University of Bath and the Tired of Cancer research team, who initially developed the Untire app. The investigators have also consulted with the Bristol Haematology and Oncology centre who will act as a recruitment site. two cancer survivors were also consulted on study methodology as well of other user experience aspects of the study design.

Conflict of interest:

The investigators are consulting with Tired of cancer (A mental health start-up company) who first developed the Untire app however the study is being independently run by the University of Bath's psychology department. Tired of Cancer are not providing any financial support / incentives for developing this study. No members of the study team are working as clinicians within the Bristol Haematology and Oncology centre.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cancer or cancer survivors (18 years and older).
* Self-reported current diagnosis or previous history of treatment for cancer (cancer survivor).
* A moderate or severe level of fatigue as measured by items 1-3 of the Brief Fatigue Inventory (BFI).
* Access to a smart phone, tablet, or iPad (Apple or Android).

Exclusion Criteria:

* Participants < 18 years of age
* Non-English language speakers
* Participants with a diagnosis of and receiving treatment for severe psychological distress (e.g. major depression, psychotic disorder, anxiety disorder, or addiction).
* Participants with a diagnosis of chronic fatigue syndrome, myalgic encephalomyelitis, or fibromyalgia.
* Previous or current us of the Untire app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The change in mean level of acceptability (as measured by the Acceptability E-scale) | From 2 weeks to final time point at 12 weeks. Participants will complete this scale at four time points (after 2 weeks, 4 weeks, 6 weeks and 12 weeks of app use).
  Acceptability E-scale has strong psychometric properties and can be useful in assessing the acceptability and usability of computerized health-related programs in oncology and other health populations.
  This is a six-item scale measuring how easy and enjoyable the app is to use, how understandable were the questions, how helpful was completing the intervention, whether the amount of time to complete the program was acceptable, and overall satisfaction with the program. This is a valid and reliable measure which has previously been used to evaluate patient perceptions of e-health interventions in an oncology setting.
  Responses are on a simple 5-point numerical scale; 1 indicates a negative and 5 indicates a positive evaluation. Scores range can range from 6-30 with higher scores indicating a higher level of acceptability. The scale will be adapted with the appropriate wording for this study.
The change in mean level of digital working alliance (as measured by the Digital working Alliance Inventory, D-WAI). | From 2 weeks to final time point at 12 weeks. Participants will complete the D-WAI at four timepoints (after 2 weeks, 4 weeks, 6 weeks and 12 weeks of app use).
  The D-WAI is a brief questionnaire used to assess digital working alliance. The 6-items are based on the successful validation of a short form of the Working Alliance Inventory (WAI-SR) comprising of the same core factors of Goals, tasks, and bond. The D-WAI has adequate internal consistency and test-retest reliability. It is a 6-item self-report questionnaire with responses rated on a seven-point Likert scale, ranging from 1 (strongly disagree) to 7 (Strongly agree).

SECONDARY OUTCOMES:
The change in mean level of fatigue (as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue, FACT-F) | From baseline to final time point at 12 weeks. Participants will complete the FACT-F at five time points (at baseline and after 2 and then again after 2 weeks (T2), 4 weeks (T4), 6 weeks (T6) and after completion of the intervention at week 12 (T12).
  This is a 40-item questionnaire which comprised of the 27-item Functional Assessment of Chronic Illness Therapy - General (FACT-G) designed to measure four domains of Health related QOL in cancer patients: Physical, social, emotional, and functional well-being. The FACT-F included an additional 13-item subscale that can be used as an independent measure of fatigue and its impact.
  The FACT-G (core subscales) has been shown to have good test-retest reliability (r=0.87) and excellent internal consistency (alphas = 0.95) on both initial and retest administrations. The fatigue subscale has independently demonstrated good test-retest reliability (r=0.90) and internal consistency (alphas = 0.93 and 0.95) on initial and test-retest administrations.
  Responses are measured on a five-point Likert scale, ranging from 0 (not at all) to 4 (very much). Scores range from 0-52 with higher scores indicating less fatigue symptoms. The measure takes 10-15 minutes to complete.
The change in mean level of quality of life (as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue, FACT-F) | From baseline to final time point at 12 weeks. Participants will complete the FACT-F at baseline, and then after 2 weeks, 4 weeks, 6 weeks and 12 weeks of app use.
  This is a 40-item questionnaire which comprised of the 27-item Functional Assessment of Chronic Illness Therapy - General (FACT-G) designed to measure four domains of Health related QOL in cancer patients: Physical, social, emotional, and functional well-being. The FACT-F included an additional 13-item subscale that can be used as an independent measure of fatigue and its impact.
  The FACT-G (core subscales) has been shown to have good test-retest reliability (r=0.87) and excellent internal consistency (alphas = 0.95) on both initial and retest administrations. The fatigue subscale has independently demonstrated good test-retest reliability (r=0.90) and internal consistency (alphas = 0.93 and 0.95) on initial and test-retest administrations.
  Responses are measured on a five-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0-108 with higher scores indicating better quality of life. The measure takes 10-15 minutes to complete.

OTHER OUTCOMES:
Brief Fatigue Inventory (BFI) | Potential participants will be asked to complete the BFI at baseline
  Items 1-3 of the Brief Fatigue Inventory will be used for eligibility screening. These three items ask participants to:
  1. Please rate their fatigue right now.
  2. Please rate their usual level of fatigue over the past 24 hours.
  3. Please rate their worst level of fatigue over the past 24 hours.
  Responses are measured on a ten-point numeric scale ranging from 0 (no fatigue) to 10 (as bad as you can imagine). In order to take part in the study participants will need to score an average composite score of ≥4 on the three items which will be considered to represent clinically meaningful fatigue. Higher scores indicate more severe fatigue.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - University Hospitals Bristol & Weston NHS Foundation Trust, Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8. doi: 10.1016/j.apnr.2009.04.003. Epub 2009 Sep 18. PMID 20974066
- [Background] Underhill ML, Hong F, Jones T, Sprunck-Harrild K, Walsh SK, Boyajian R, Berry DL, Partridge A. Feasibility and Acceptability of a Web Site to Promote Survivorship Care in Survivors of Hodgkin Disease. JCO Clin Cancer Inform. 2017 Nov;1:1-10. doi: 10.1200/CCI.17.00012. PMID 30657382
- [Background] Henson P, Wisniewski H, Hollis C, Keshavan M, Torous J. Digital mental health apps and the therapeutic alliance: initial review. BJPsych Open. 2019 Jan;5(1):e15. doi: 10.1192/bjo.2018.86. PMID 30762511
- [Background] Goldberg SB, Baldwin SA, Riordan KM, Torous J, Dahl CJ, Davidson RJ, Hirshberg MJ. Alliance With an Unguided Smartphone App: Validation of the Digital Working Alliance Inventory. Assessment. 2022 Sep;29(6):1331-1345. doi: 10.1177/10731911211015310. Epub 2021 May 18. PMID 34000843
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Spahrkas SS, Looijmans A, Sanderman R, Hagedoorn M. How does the Untire app alleviate cancer-related fatigue? A longitudinal mediation analysis. Psychooncology. 2022 Jun;31(6):970-977. doi: 10.1002/pon.5886. Epub 2022 Jan 27. PMID 35060222
- [Background] Spahrkas SS, Looijmans A, Sanderman R, Hagedoorn M. Beating Cancer-Related Fatigue With the Untire Mobile App: Protocol for a Waiting List Randomized Controlled Trial. JMIR Res Protoc. 2020 Feb 14;9(2):e15969. doi: 10.2196/15969. PMID 32130185

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05891431/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05891431/ICF_001.pdf